CLINICAL TRIAL: NCT01859390
Title: A Multi-Center, Randomized, Controlled, Double-Blind Study of the Effects of an Antioxidant-Enriched Multivitamin Supplement on Inflammation and Oxidative Stress in Cystic Fibrosis Patients
Brief Title: Effects of an Antioxidant-Enriched Multivitamin Supplement on Inflammation and Oxidative Stress in Cystic Fibrosis
Acronym: AquADEKs-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Yasoo Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-1557; AQUADEK12K1 (Other: Medic)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Cystic Fibrosis
Keywords: Antioxidants; Vitamins; Inflammation; Oxidative stress
MeSH Terms: conditions — Cystic Fibrosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AquADEKs-2 (Experimental): Two control multivitamin softgel capsules will be taken orally on a once daily basis with pancreatic enzymes and a glass of milk or fat-containing meal for 4 weeks for the screening run in period. For those subjects randomized to the AquADEKs-2 arm, two AquADEKs-2 softgel capsules will be taken orally on a once daily basis with pancreatic enzymes and a glass of milk or fat-containing meal for 16 weeks.
  Interventions: Drug: AquADEKs-2; Dietary Supplement: control multivitamin
- Control multivitamin (Active Comparator): Two control multivitamin softgel capsules will be taken orally on a once daily basis with pancreatic enzymes and a glass of milk or fat-containing meal for 4 weeks for the screening run in period for all participants and for 16 weeks for those randomized to this comparative therapy.
  Interventions: Dietary Supplement: control multivitamin

INTERVENTIONS:
Drug: AquADEKs-2 — AquADEKs-2 contains standard amounts of fat-soluble vitamins (A, D, E, K) that are contained in typical CF multivitamin supplements plus several antioxidants including beta-carotene, mixed tocopherols (different forms of vitamin E), coenzyme Q10 (CoQ10), mixed carotenoids (lutein, lycopene and zeaxanthin), and the minerals zinc and selenium.
  Other Names: Antioxidant-enriched multivitamin supplement
  Arms: AquADEKs-2
Dietary Supplement: control multivitamin — The control multivitamin contains standard (standard for CF multivitamin supplements) amounts of vitamins A, B, D, E, and K without added antioxidants.

SUMMARY:
The purpose of this study will be to evaluate the effects of a modified formulation of AquADEKs (AquADEKs-2) on markers of inflammation, antioxidant levels and oxidative stress.

Cystic Fibrosis (CF) is a disease that affects the organs in the body such as the lungs. Some of the damage to the lungs of CF patients may be caused by something called oxidant/antioxidant imbalance and oxidative stress.

Oxidation in the body is kind of what happens to an apple when it turns brown after being cut. And, just as a squeeze of lemon juice stops the oxidation of an apple, antioxidants can stop the rusting (or damage) inside our bodies by unstable oxygen molecules called free radicals. Free radicals can help fight off bacteria and viruses but too many of them do damage instead. Our bodies need antioxidants to keep things in balance so we have the right amount of free radicals.

Many CF patients also have trouble digesting food and absorbing nutrients like vitamins. Many of the vitamins we rely on are antioxidants, like vitamins A, D, E, K and beta-carotene. In some people with CF, even though they take multivitamins and pancreatic enzymes, they still have low amounts of antioxidants. The investigators are looking to see if taking more vitamins and antioxidants will help CF patients.

AquADEKs-2 is an investigational new drug (a drug that has not received approval by the Food and Drug Administration [FDA]). This research study is being done with the AquADEKs-2 compared to a control multivitamin. The study drug, AquADEKs-2 contains standard amounts of fat-soluble vitamins (A, D, E, K) that are contained in typical CF multivitamin supplements plus several antioxidants including beta-carotene, mixed tocopherols (different forms of vitamin E), coenzyme Q10 (CoQ10), mixed carotenoids (lutein, lycopene and zeaxanthin), and the minerals zinc and selenium. The control multivitamin contains standard amounts of vitamins A, B, D, E, and K without additional antioxidant supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥10 years of age
* Documentation of a Cystic Fibrosis (CF) diagnosis as evidenced by 1 or more clinical features consistent with the CF phenotype and 1 or more of the following criteria:

  * Sweat chloride equal to or greater than 60 milliequivalent (mEq/L) by quantitative pilocarpine iontophoresis test (QPIT)
  * 2 well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
* Pancreatic insufficiency documented by having a spot fecal elastase-1 (FE-1) ≤ 100μg/g in a stool sample done either historically or at the screening visit
* Clinically stable with no significant changes in health status within 2 weeks prior to randomization
* Forced expiratory volume over one second (FEV1) ≥ 40 and ≤ 100% of predicted for age based on the Wang (males < 18 years,females < 16 years) or Hankinson (males ≥ 18 years, females ≥ 16 years) standardized equations at the screening visit
* Weight ≥ 30 kg at the screening visit
* Able to perform repeatable, consistent efforts in pulmonary function testing
* Able to tolerate sputum induction with 3% hypertonic saline and to expectorate with induction
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative
* Ability to swallow softgel capsules

Exclusion Criteria:

* Subjects being treated with ivacaftor (Kalydeco™)
* Liver enzymes aspartate aminotransferase (AST), alanine aminotransferase (ALT), or gamma-glutamyl transferase (GGT) > 3 times the upper limits of normal at the screening visit
* Use of antibiotics (oral, iv, and/or inhaled) for acute respiratory symptoms within 2 weeks prior to randomization
* Active treatment for allergic bronchopulmonary aspergillosis (ABPA)
* Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone/day or 20 mg prednisone every other day
* Active treatment for nontuberculous mycobacterial (NTM) infection
* Initiation of any new chronic therapy (e.g., ibuprofen, Pulmozyme®, hypertonic saline,azithromycin,Tobramycin Inhalation solution (TOBI®), Cayston® within 8 weeks prior to randomization
* Unwilling to discontinue current oral vitamin and antioxidant supplementation (e.g.,AquADEKs®, another source of β-carotene, vitamin A, vitamin E or tocopherols,vitamins D or K, n-acetylcysteine, glutathione, CoQ10, other over-the-counter antioxidant) for the duration of the study
* Use of vitamins (other than control vitamin) or antioxidants within 4 weeks prior to randomization
* Daily use of > 2 cans of Boost or Pulmocare dietary supplement formulas
* Known hypersensitivity to oral AquADEKs®
* For women of child bearing potential:

  1. positive pregnancy test at Visit 1 or at Visit 2, or
  2. lactating or
  3. unwilling to practice a medically acceptable form of contraception (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent)
* Subject unlikely to complete the study as determined by the Investigator
* Any condition that the Investigator believes would interfere with the intent of this study or would make participation not in the best interest of the subject
* Use of investigational therapies within 4 weeks prior to randomization
* Current tobacco smoker
* Current use of anticoagulant medications
* Severe malnutrition based either on having a BMI less than the 5th percentile for subjects < 18 years of age or a body mass index (BMI) less than 18 kg/m2 for subjects > 18 years of age.
* Subjects with poorly controlled CF-related diabetes on active insulin therapy, defined as having a Glycosylated Hemoglobin (HgbA1c) ≥ 7.5% at the most recent historic evaluation of HgbA1c

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sagel, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (15):
- United States (15):
  - University Medical Center, Tucson, Arizona
  - Children's Hospital Colorado, Aurora, Colorado
  - The Nemours Children's Clinic, Orlando, Florida
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Wisconsin Hospital Center, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sagel SD, Sontag MK, Anthony MM, Emmett P, Papas KA. Effect of an antioxidant-rich multivitamin supplement in cystic fibrosis. J Cyst Fibros. 2011 Jan;10(1):31-6. doi: 10.1016/j.jcf.2010.09.005. Epub 2010 Oct 20. PMID 20961818
- [Background] Papas KA, Sontag MK, Pardee C, Sokol RJ, Sagel SD, Accurso FJ, Wagener JS. A pilot study on the safety and efficacy of a novel antioxidant rich formulation in patients with cystic fibrosis. J Cyst Fibros. 2008 Jan;7(1):60-7. doi: 10.1016/j.jcf.2007.05.001. Epub 2007 Jun 13. PMID 17569601
- [Derived] Jain R, Baines A, Khan U, Wagner BD, Sagel SD. Evaluation of airway and circulating inflammatory biomarkers for cystic fibrosis drug development. J Cyst Fibros. 2021 Jan;20(1):50-56. doi: 10.1016/j.jcf.2020.06.017. Epub 2020 Jul 1. PMID 32622665
- [Derived] Sagel SD, Khan U, Jain R, Graff G, Daines CL, Dunitz JM, Borowitz D, Orenstein DM, Abdulhamid I, Noe J, Clancy JP, Slovis B, Rock MJ, McCoy KS, Strausbaugh S, Livingston FR, Papas KA, Shaffer ML. Effects of an Antioxidant-enriched Multivitamin in Cystic Fibrosis. A Randomized, Controlled, Multicenter Clinical Trial. Am J Respir Crit Care Med. 2018 Sep 1;198(5):639-647. doi: 10.1164/rccm.201801-0105OC. PMID 29688760

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AquADEKs-2 | Control Multivitamin
Started (Randomized) | 36 | 37
Withdrawals (Participants can withdraw anytime prior to their Week 18 follow-up visit.) | 2 | 2
Completed (Based on availability of Week 16 sputum myeloperoxidase (MPO) measurement (primary endpoint)) | 35 | 30
Not Completed | 1 | 7
Not completed — Insufficient Sputum Collected | 1 | 3
Not completed — Sample Missing Collection Date | 0 | 1
Not completed — Tube Cracked | 0 | 2
Not completed — Shipment Error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AquADEKs-2 | Control Multivitamin | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (8.9) | 22.9 (9.5) | 22.6 (9.1)
Age, Customized [Count of Participants; unit: Participants] — Age Category (10-18 years, 18-30 years, 30+ years)
  Participants
    Age >=10 - <18 yrs | 13 | 16 | 29
    Age >=18 - <30 yrs | 17 | 11 | 28
    Age >30 yrs | 6 | 10 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 16 | 17 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 34 | 30 | 64
  Race/Ethnicity: Hispanic | 1 | 5 | 6
  Race/Ethnicity: African-American | 1 | 1 | 2
  Race/Ethnicity: Unknown/Other | 0 | 1 | 1
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants]
  Delta F508 Homozygous | 23 | 16 | 39
  Delta F508 Heterozygous | 9 | 18 | 27
  Other | 3 | 3 | 6
  Not Identified | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Sputum Myeloperoxidase (MPO) Level
Description: The primary outcome is the difference in 16 week mean change in log10 sputum myeloperoxidase levels between the AquADEKs-2 arm and the Control Multivitamin arm.
Time Frame: Baseline (Visit 2) to Week 16 (Visit 4)
Measure: Mean (Standard Deviation); unit: log10 (ng/mL)
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 35 | 30
log10 (ng/mL) | -0.10 (0.67) | 0.03 (0.76)
Statistical Analysis 1: Comparison: AquADEKs-2 vs Control Multivitamin; Two-sample T-test; Test type: Superiority; p = 0.460, t-test, 2 sided; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.49 to 0.22]
Statistical Analysis 2: Comparison: AquADEKs-2 vs Control Multivitamin; Test type: Superiority; p = 0.325, Regression, Linear; Mean Difference (Final Values) = -0.170, 95% CI 2-sided [-0.513 to 0.173] — Regression Model predictors include: AquADEKs-2 arm, Age >=18 years, Sex, Screening FEV1%Predicted >70%, Chronic use of Inhaled Antibiotics and Azithromycin. The estimated value is the mean difference between groups for 16 week change in log10 MPO

2. Secondary Outcome: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Incidence is defined as the number and percentage of participants with at least one event over the 18 week follow-up period.
Time Frame: 18 weeks follow up
Measure: Count of Participants; unit: Participants
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 36 | 37
Participants
  Incidence of AEs | 33 | 34
  Incidence of SAEs | 8 | 13
Statistical Analysis 1: Comparison: AquADEKs-2 vs Control Multivitamin; Test type: Superiority; p = 0.302, Fisher Exact; Difference in Proportions-SAE incidence = -12.9, 95% CI 2-sided [-32.1 to 7.8]

3. Secondary Outcome: Rate of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Rate is defined as the number of events per participant follow-up week.
Time Frame: 18 weeks follow up
Measure: Number; unit: events per participant-week
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 36 | 37
events per participant-week
  Number of AEs per participant week | 0.34 | 0.37
  Number of SAEs per participant week | 0.04 | 0.05
Statistical Analysis 1: Comparison: AquADEKs-2 vs Control Multivitamin; Rate Ratio for Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in weeks. The total number of follow-up weeks in the AquADEKs-2 group was 642 and in the Control group was 639; Test type: Superiority; p = 0.486, Poisson Model; Rate Ratio = 0.94, 95% CI 2-sided [0.78 to 1.13]
Statistical Analysis 2: Comparison: AquADEKs-2 vs Control Multivitamin; Test type: Superiority — Rate Ratio for Serious Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in weeks. The total number of follow-up weeks in the AquADEKs-2 group was 642 and in the Control group was 639; p = 0.269, Poisson Regression; Rate Ratio = 0.74, 95% CI 2-sided [0.43 to 1.26]

4. Secondary Outcome: Change in Lung Function
Description: Absolute Change in Forced Expiratory Volume over one second (FEV1) % predicted between Baseline and Week 16. Global Lung Initiative equations were used to calculate FEV1 %predicted.
Time Frame: Baseline (Visit 2) to Week 16
Population: This population includes participants who did not complete the study (i.e., did not have a final analyzable sputum sample) but did have a final lung function assessment.
Measure: Mean (Standard Deviation); unit: FEV1 %Predicted
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 34 | 35
FEV1 %Predicted | -0.76 (8.00) | -2.20 (7.53)
Statistical Analysis 1: Comparison: Control Multivitamin; Test type: Superiority — Two sample T-test; p = 0.4463, t-test, 2 sided; Median Difference (Final Values) = 1.43, 95% CI 2-sided [-2.30 to 5.16]

5. Secondary Outcome: Change in Growth Endpoints
Description: Absolute change in Body Mass Index (BMI) (kg/m^2) between Baseline and Week 16.
Time Frame: Baseline (Visit 2) to Week 16
Population: This population includes participants who did not complete the study (i.e., did not have a final analyzable sputum sample) but did have final height and weight assessments.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 34 | 34
kg/m^2 | 0.16 (0.68) | 0.13 (0.96)
Statistical Analysis 1: Comparison: AquADEKs-2 vs Control Multivitamin; Test type: Superiority; p = 0.8623, t-test, 2 sided; Median Difference (Final Values) = 0.04, 95% CI 2-sided [-0.37 to 0.44]

6. Secondary Outcome: Time to First Pulmonary Exacerbation
Description: Median time to first pulmonary exacerbation (PEx) between baseline (Visit 2) and end of follow up (Week 18)
Time Frame: Baseline (Visit 2) to end of follow up (Week 18)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 36 | 37
days | 102 [78 to NA] — The upper bound of the confidence interval could not be computed due to the distribution of events in the AquADEKs-2 arm. | 96 [35 to 125]
Statistical Analysis 1: Comparison: AquADEKs-2 vs Control Multivitamin; Test type: Superiority; p = 0.0534, Regression, Cox — Not adjusted for multiple comparisons. Alpha at 0.05; Cox Proportional Hazard = 0.536, 95% CI 2-sided [0.284 to 1.009] — Cox model parameters include: AquADEKs-2 arm, Age >=18 years, Sex, Screening FEV1 % Predicted >70%, Chronic use of Inhaled Antibiotics and Azithromycin. The parameter of interest is the Hazard Ratio comparing the AquADEKs-2 arm to the control arm

7. Secondary Outcome: Number of Pulmonary Exacerbations
Description: The total number of PEx between baseline (Visit 2) and end of follow up (Week 18).
Time Frame: Baseline (Visit 2) to end of follow up (Week 18)
Measure: Number; unit: Pulmonary Exacerbations
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 36 | 37
Pulmonary Exacerbations | 28 | 39
Statistical Analysis 1: Comparison: AquADEKs-2 vs Control Multivitamin; Rate Ratio for PEx calculated using Poisson Regression with an offset for the log of follow-up time in months. The total number of follow-up months in the AquADEKs-2 group was 148 and in the Control group was 147; Test type: Superiority; p = 0.1731, Poisson Model; Rate Ratio = 0.72, 95% CI 2-sided [0.44 to 1.16]

8. Secondary Outcome: Number of Participants With Pulmonary Exacerbations
Description: Number (%) with at least one protocol-defined PEx between baseline (Visit 2) and end of follow up (Week 18).
Time Frame: Baseline (Visit 2) to end of follow up (Week 18)
Measure: Count of Participants; unit: Participants
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 36 | 37
Participants | 19 | 25
Statistical Analysis 1: Comparison: AquADEKs-2 vs Control Multivitamin; Test type: Superiority — Difference in Proportions; p = 0.2363, Fisher Exact — Not adjusted for multiple comparisons. Alpha at 0.05; Mean Difference (Final Values) = -14.8, 95% CI 2-sided [-35.1 to 7.4]

9. Secondary Outcome: Number of Participants Hospitalized
Description: Number (%) of participants with at least one hospitalization between Baseline (Visit 2) and end of follow up (Week 18).
Time Frame: Baseline (Visit 2) to end of followup (Week 18)
Measure: Count of Participants; unit: Participants
Arm/Group | AquADEKs-2 | Control Multivitamin
Number analyzed (Participants) | 36 | 37
Participants | 7 | 13
Statistical Analysis 1: Comparison: Control Multivitamin; Test type: Superiority — Difference in Proportions; p = 0.1900, Fisher Exact; Median Difference (Final Values) = -15.7, 95% CI 2-sided [-34.5 to 4.8]

ADVERSE EVENTS:
Time Frame: Participant adverse event data was collected for the 4 months that subjects were on study drug.
Arm/Group | AquADEKs-2 | Control Multivitamin
Serious Adverse Events (participants affected / at risk) | 8/36 | 13/37
Other Adverse Events (participants affected / at risk) | 33/36 | 34/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AquADEKs-2 (N=36) | Control Multivitamin (N=37)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1)
Chest X-ray abnormal (Investigations) | 0 (0) | 1 (2)
Forced expiratory volume decreased (Investigations) | 2 (2) | 1 (1)
Pulmonary function test decreased (Investigations) | 2 (2) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AquADEKs-2 (N=36) | Control Multivitamin (N=37)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 8 (11)
Constipation (Gastrointestinal disorders) | 1 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (4) | 5 (7)
Pyrexia (General disorders) | 2 (2) | 5 (6)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Forced expiratory volume decreased (Investigations) | 2 (3) | 1 (1)
Pseudomonas test positive (Investigations) | 0 (0) | 2 (2)
Pulmonary function test decreased (Investigations) | 6 (9) | 9 (10)
Weight decreased (Investigations) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 4 (7) | 5 (5)
Sinus headache (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Decreased activity (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (30) | 19 (30)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 10 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
We did not meet the complete enrollment of 80 subjects due to the expiration dates of the antioxidant-enriched and control multivitamins produced for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No